CLINICAL TRIAL: NCT01865331
Title: A Randomised, Double-blind, Placebo-controlled, Single-dose, Parallel Group Trial With Insulin 454 and SIAM 50 in Healthy Male Japanese Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic and Pharmacodynamic Characteristics of Explorative Formulations of Insulin Degludec and IDegAsp 50 in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1788; 2006-002615-26 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose, insulin degludec (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- Medium dose, insulin degludec (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- High dose, insulin degludec (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- IDegAsp 50 (Experimental)
  Interventions: Drug: placebo; Drug: insulin degludec/insulin aspart 50

INTERVENTIONS:
Drug: insulin degludec — Single dose administered subcutaneously (s.c., under the skin).
  Arms: High dose, insulin degludec; Low dose, insulin degludec; Medium dose, insulin degludec
Drug: placebo — Administered subcutaneously (s.c., under the skin)
Drug: insulin degludec/insulin aspart 50 — Single dose of IDegAsp 50 administered subcutaneously (s.c., under the skin)
  Arms: IDegAsp 50

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate safety, tolerability and pharmacokinetic (the exposure of the trial drug in the body) and pharmacodynamic (the effect of the investigated drug on the body) characteristics of insulin degludec (insulin 454) and insulin degludec/insulin aspart (IDegAsp) 50 - formerly SIAM), both explorative formulations, not similar to the proposed commercial formulation, in healthy male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese passport holder
* Japanese-born parents
* Body mass index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)
* Fasting blood glucose of below or equal to 6 mmol/L
* Healthy male subjects, who are considered to be generally healthy based on an assessment of medical history, physical examination and clinical laboratory data at screening, as assessment of medical history, physical exjudged by the Investigator

Exclusion Criteria:

* The receipt of any investigational drug within 3 months prior to this trial
* Subjects with a history of significant multiple drug allergies or with a known allergy to the trialproduct or any medicine chemically related to the trial product, as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | From dosing visit and until follow-up 7-21 days after last dosing visit

SECONDARY OUTCOMES:
Area under the serum insulin concentration curve | 0-96 hours after dosing
Area under the glucose infusion rate curve | 0-24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com